CLINICAL TRIAL: NCT02445560
Title: The Effects of a High Protein Diet on Microbiota, Gastrointestinal Function, Wellness and the Potential Mitigating Effects of a Multi-strain Probiotic, Prebiotic, and Synbiotic: a Randomized, Double-blinded Crossover Study in Older Women.
Brief Title: The Effects of a High Protein Diet on Microbiota, Gastrointestinal Function and Wellness in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201400955
Record Dates: First submitted 2015-04-06; First posted 2015-05-15 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Aging
Keywords: probiotics; prebiotics; high protein diet; microbiota
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Probiotic capsule and Fiber sachet (Experimental): Participants will be randomly assigned to receive all of the following in random order: a probiotic capsule and fiber sachet daily for 2-weeks, a probiotic capsule and placebo sachet for 2-weeks, a fiber sachet and placebo capsule for 2-weeks, and placebo capsule and placebo sachet for 2-weeks. Each treatment period is separated by a 2-week washout. During each treatment period, in addition to consuming a probiotic capsule or placebo and/or a fiber sachet or placebo sachet participants will be on a controlled higher protein diet.
  Interventions: Dietary Supplement: Probiotic capsule and Placebo sachet; Dietary Supplement: Placebo capsule and Fiber Sachet; Dietary Supplement: Placebo capsule and Placebo sachet
- Probiotic capsule and Placebo sachet (Experimental): Participants will be randomly assigned to receive all of the following in random order: a probiotic capsule and fiber sachet daily for 2-weeks, a probiotic capsule and placebo sachet for 2-weeks, a fiber sachet and placebo capsule for 2-weeks, and placebo capsule and placebo sachet for 2-weeks. Each treatment period is separated by a 2-week washout. During each treatment period, in addition to consuming a probiotic capsule or placebo and/or a fiber sachet or placebo sachet participants will be on a controlled higher protein diet.
  Interventions: Dietary Supplement: Probiotic capsule and Fiber Sachet; Dietary Supplement: Placebo capsule and Fiber Sachet; Dietary Supplement: Placebo capsule and Placebo sachet
- Placebo capsule and Fiber sachet (Experimental): Participants will be randomly assigned to receive all of the following in random order: a probiotic capsule and fiber sachet daily for 2-weeks, a probiotic capsule and placebo sachet for 2-weeks, a fiber sachet and placebo capsule for 2-weeks, and placebo capsule and placebo sachet for 2-weeks. Each treatment period is separated by a 2-week washout. During each treatment period, in addition to consuming a probiotic capsule or placebo and/or a fiber sachet or placebo sachet participants will be on a controlled higher protein diet.
  Interventions: Dietary Supplement: Probiotic capsule and Fiber Sachet; Dietary Supplement: Probiotic capsule and Placebo sachet; Dietary Supplement: Placebo capsule and Placebo sachet
- Placebo capsule and Placebo sachet (Placebo Comparator): Participants will be randomly assigned to receive all of the following in random order: a probiotic capsule and fiber sachet daily for 2-weeks, a probiotic capsule and placebo sachet for 2-weeks, a fiber sachet and placebo capsule for 2-weeks, and placebo capsule and placebo sachet for 2-weeks. Each treatment period is separated by a 2-week washout. During each treatment period, in addition to consuming a probiotic capsule or placebo and/or a fiber sachet or placebo sachet participants will be on a controlled higher protein diet.
  Interventions: Dietary Supplement: Probiotic capsule and Fiber Sachet; Dietary Supplement: Probiotic capsule and Placebo sachet; Dietary Supplement: Placebo capsule and Fiber Sachet

INTERVENTIONS:
Dietary Supplement: Probiotic capsule and Fiber Sachet — A probiotic capsule and fiber sachet will be consumed daily for 2-weeks. The probiotic capsule contains a mixture of Bifidobacterium bifidum, Bifidobacterium breve, Bifidobacterium longum, Lactobacillus acidophilus and Lactobacillus plantarum. The fiber sachet consists of 5 g of chicory root fiber.
  During the treatment period, in addition to consuming the probiotic capsule and fiber sachet participants will consume a controlled diet consisting of foods that provide an average of approximately 2 g/kg/day of protein.
  Arms: Placebo capsule and Fiber sachet; Placebo capsule and Placebo sachet; Probiotic capsule and Placebo sachet
Dietary Supplement: Probiotic capsule and Placebo sachet — A probiotic capsule and placebo sachet will be consumed daily for 2-weeks. The probiotic capsule contains a mixture of Bifidobacterium bifidum, Bifidobacterium breve, Bifidobacterium longum, Lactobacillus acidophilus and Lactobacillus plantarum. The placebo sachet consists of 5 g of maltodextrin.
  During the treatment period, in addition to consuming the probiotic capsule and placebo sachet participants will consume a controlled diet consisting of foods that provide an average of approximately 2 g/kg/day of protein.
  Arms: Placebo capsule and Fiber sachet; Placebo capsule and Placebo sachet; Probiotic capsule and Fiber sachet
Dietary Supplement: Placebo capsule and Fiber Sachet — A placebo capsule and fiber sachet will be consumed daily for 2-weeks. The placebo capsule will contain potato starch, magnesium stearate and ascorbic acid. The fiber sachet consists of 5 g of chicory root fiber.
  During the treatment period, in addition to consuming the placebo capsule and fiber sachet participants will consume a controlled diet consisting of foods that provide an average of approximately 2 g/kg/day of protein.
  Arms: Placebo capsule and Placebo sachet; Probiotic capsule and Fiber sachet; Probiotic capsule and Placebo sachet
Dietary Supplement: Placebo capsule and Placebo sachet — A placebo capsule and placebo sachet will be consumed daily for 2-weeks. The placebo capsule will contain potato starch, magnesium stearate and ascorbic acid. The fiber sachet consists of 5 g of maltodextrin.
  During the treatment period, in addition to consuming the placebo capsule and placebo sachet participants will consume a controlled diet consisting of foods that provide an average of approximately 2 g/kg/day of protein.
  Arms: Placebo capsule and Fiber sachet; Probiotic capsule and Fiber sachet; Probiotic capsule and Placebo sachet

SUMMARY:
The purpose of the proposed study is to determine the effects of consuming a high protein diet on fecal microbial communities, gastrointestinal function and symptoms, and general wellness in older adults.

DETAILED DESCRIPTION:
Older women will be randomized to a 18-week crossover study design. During each treatment period participants will be provided with a weight maintenance diet providing approximately 2 g/kg/day of protein.

Following a two-week baseline and in random order will have the following diets assigned:

The participants will be provided with a weight maintenance, high protein diet for two weeks, then for two-weeks will resume their normal diet;

The participants will come back into clinic and for the next two weeks to receive a high protein diet with a multi-strain probiotic for two weeks, then for two-weeks will resume their normal diet;

The participants will come back into clinic and for the next two weeks will receive a high protein diet with a prebiotic, then for two-weeks will resume their normal diet;

The participants will come back into clinic and for the next two weeks will receive a high protein diet with the synbiotic combination. then for two-weeks will resume their normal diet

Participants and researchers will be blinded for each treatment period (participants will receive a probiotic or placebo capsule, and a prebiotic or placebo sachet).

The following will be performed during the clinic visits: Questionnaires will assess quality of life (QoL), wellness, gastrointestinal symptoms, bowel movement frequency, and compliance. Hand-grip strength will be measured. Blood and urine samples will be collected at baseline and at weeks 2, 6,10 and 14. Stool samples will be collected at baseline and at weeks 2, 4, 6, 8,10, 12, 14 and 16.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study you must

* be a woman 65 years of age or older
* be willing to complete daily and weekly questionnaires
* be willing to wear a SenseWear Pro Armband (BodyMedia, Inc.) to monitor energy expenditure and establish dietary energy needs
* be willing to provide blood samples, stool samples, and urine samples throughout the course of the study
* be willing to discontinue prebiotics, probiotics and/or any fiber supplements for the duration of the study
* be willing to consume the provided diet for the designated 8 weeks of the study
* are willing to report and maintain their usual alcohol intake throughout the study
* are able to take foods, study fiber, probiotic, and placebo without the aid of another person
* able to attend all scheduled study appointments for the duration of the study
* have a usual protein intake consistent with United States' population as assessed by dietary analysis
* have a usual fiber intake consistent with United States' population as assessed by dietary analysis
* be willing to provide a social security number to receive study payment.

Exclusion Criteria:

To participate in the study you must NOT

* have a physician-diagnosed gastrointestinal disease or condition (such as ulcerative colitis, Crohn's disease, gastroparesis, peptic ulcer disease, cancer, celiac disease, short bowel disease, ileostomy)
* have had or are currently being treated for any known illnesses or conditions that may impact perceived health such as HIV/AIDS, immune modulating diseases (autoimmune, hepatitis, cancer, etc.), diabetes or chronic kidney disease
* be a vegetarian
* have any known food allergies or dietary restrictions
* be currently taking medication for constipation or diarrhea
* have taken antibiotics within the past 2 months
* be a current smoker
* be planning on loosing/gaining weight during the next 6 months
* typically consume no more than one alcoholic beverage per day
* have a BMI greater than 30

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Microbiota Studies (recovery) | Change from Baseline at Week 2,4,6,8,10,12,14,16
  Change in the concentrations of the probiotic strains in the stools will be measured with strain specific deoxyribonucleic acid (DNA) (or antibodies) in fecal samples (e.g. quantitative polymerase chain reaction (qPCR), flow cytometry).
Microbiota Studies (overall composition) | Change from Baseline at Week 2,4,6,8,10,12,14,16
  Effects of the probiotic interventions on overall microbiota composition (e.g. 454 16S rRNA (ribosomal ribonucleic acid) sequencing) will also be measured.

SECONDARY OUTCOMES:
Digestive Health (Gastrointestinal Symptom Rating Scale ) | Change from Baseline at Week 1,2,3,4,5,6,7,8,9,10,11,12,13,14,15,16,17,18
  Measured by gastrointestinal symptoms (gas, bloating, diarrhea, etc.) assessed using the weekly Gastrointestinal Symptom Rating Scale (GSRS).
Digestive Health (Bristol Stool Scale) | Change from Baseline at Week 1,2,3,4,5,6,7,8,9,10,11,12,13,14,15,16,17,18
  Measured by gastrointestinal symptoms (gas, bloating, diarrhea, etc.) assessed using a daily questionnaire. The daily questionnaire will include questions regarding symptoms and the Bristol Stool Scale (stool form and transit).
Blood Analysis (metabolic) | Change from Baseline at Weeks 2,6,10,14
  Measured by comprehensive Metabolic Panel
Blood Analysis (lipids) | Change from Baseline at Weeks 2,6,10,14
  Measured by Lipid Panel
Blood Analysis (inflammation) | Change from Baseline at Weeks 2,6,10,14
  Measured by Inflammatory markers
Blood Analysis (blood count) | Change from Baseline at Weeks 2,6,10,14
  Measured by Complete Blood Count (CBC)
Blood Analysis (signalling) | Change from Baseline at Weeks 2,6,10,14
  Measured by (mammalian target of rapamycin) mTOR
Blood Analysis (regulation) | Change from Baseline at Weeks 2,6,10,14
  Measured by insulin-like growth factor 1 (IGF-1)
Blood Analysis (proteolysis) | Change from Baseline at Weeks 2,6,10,14
  Measured by total p-cresol
General Wellness | Day 1 through 126
  Individual reporting of antibiotic usage, visits to a physician, etc.
Proteolytic Activity | Change from Baseline at Weeks 2,6,10,14
  Measured by urinary p-cresol, indoxyl sulfate and urine urea nitrogen (UUN)
Measures of Quality of Life (QoL) | Change from Baseline at Weeks 2,6,10,14
  QoL questionnaire (domains such as physical functioning, general health, bodily pain, vitality, social functioning), questionnaire to assess frailty, and hand grip strength
Measures of Well-being (frailty) | Change from Baseline at Weeks 2,6,10,14
  Questionnaire to assess frailty
Measures of Well-being (hand grip) | Change from Baseline at Weeks 2,6,10,14
  Hand grip strength will be measured
Acceptability of the Diet | Day 1 through 126
  Acceptability will be measured using the daily questionnaire and participant compliance recordings/logs of any unconsumed foods during treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Dahl, PhD, RD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Food Science and Human Nutrition Department, Gainesville, Florida
  - UF/IFAS Extension Office Marion County, Ocala, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ford AL, Nagulesapillai V, Piano A, Auger J, Girard SA, Christman M, Tompkins TA, Dahl WJ. Microbiota Stability and Gastrointestinal Tolerance in Response to a High-Protein Diet with and without a Prebiotic, Probiotic, and Synbiotic: A Randomized, Double-Blind, Placebo-Controlled Trial in Older Women. J Acad Nutr Diet. 2020 Apr;120(4):500-516.e10. doi: 10.1016/j.jand.2019.12.009. PMID 32199523